# A Phase 1, Randomized, 2-Period, 2-Sequence, Cross-over Study to Determine the Effect of ALXN1840 on the Metabolism of a CYP2CP Substrate in Healthy Participants

**Unique Protocol ID:** ALXN1840-HV-105

NCT Number: NCT04526197

**Date of SAP:** 04 September 2020

# Alexion Pharmaceuticals, Inc.

# **ALXN1840-HV-105**

A Phase 1, Randomized, 2-Period, 2-Sequence, Cross-over Study to Determine the Effect of ALXN1840 on the Metabolism of a CYP2C9 Substrate in Healthy Participants

04Sep2020

Final Statistical Analysis Plan

Version 1.0

Prepared by:

PPD 3900 Paramount Parkway Morrisville, NC 27560 USA

Alexion 

# **TABLE OF CONTENTS**

| LIST | OF ABBREVIATIONS | 4 |
|---|---|---|
| 1. | INTRODUCTION | 6 |
| 2. | OBJECTIVES | 6 |
| 2.1.<br>2.2. | | |
| 3. | INVESTIGATIONAL PLAN | 6 |
| | | 8<br>8<br>8 |
| <b>4.</b> 4.1. | | |
| 4.2.<br>4.3.<br>4.4.<br>4.4. | | 10<br>10<br>11<br><i>11</i> |
| 5. | PARTICIPANT DISPOSITION | 11 |
| 5.1.<br>5.2. | | |
| 6. | DEMOGRAPHICS AND BASELINE CHARACTERISTICS | 12 |
| 6.1.<br>6.2.<br>6.3.<br>6.4.<br>6.5. | Urine Alcohol and Drug screen Medical History Inclusion and Exclusion Criteria | 12<br>12<br>13 |
| 7. | TREATMENTS AND MEDICATIONS | 13 |
| 7.1.<br>7.2.<br>7.3. | PRIOR AND CONCOMITANT MEDICATIONS NON-PHARMACOLOGIC THERAPIES AND PROCEDURES STUDY TREATMENTS | 13 |
| 8. | SAFETY ANALYSIS | 14 |
| 8.1.<br>8 | ADVERSE EVENTS | |

| 8 | 1.2. Relationship of Adverse Events to Study Drug | 15 |
|------|-------------------------------------------------------|----|
| 8.1 | 1.3. Intensity of Adverse Event | |
| 8 | 1.4. Serious Adverse Events | 16 |
| 8.1 | 1.5. Adverse Events Leading to drug withdrawal | 16 |
| 8.2. | CLINICAL LABORATORY EVALUATIONS | 16 |
| 8.2 | 2.1. Chemistry | 17 |
| 8.2 | 2.2. Hematology | 17 |
| 8.2 | 2.3. Coagulation | 17 |
| 8.2 | 2.4. Urinalysis | 17 |
| 8.3. | VITAL SIGN MEASUREMENTS | 17 |
| 8.4. | PHYSICAL EXAMINATION | 18 |
| 8.5. | Electrocardiogram | 18 |
| 8.6. | OTHER SAFETY DATA | 18 |
| 8.0 | 6.1. Liver Function Results | 18 |
| 8.0 | 6.2. Serology | 18 |
| 8.6 | 6.3. Pregnancy Test | 19 |
| 8.0 | 6.4. Follicle Stimulating Hormone | 19 |
| 8.0 | 6.5. Discussion/documentation of contraception method | 19 |
| 8.0 | 6.6. Retained Sample | 19 |
| 9. | PHARMACOKINETICS AND PHARMACODYNAMIC ANALYSIS | 19 |
| 9.1. | PHARMACOKINETIC SAMPLING | 19 |
| 9.2. | | |
| 9.3. | | |
| 9.4. | PHARMACOKINETIC PARAMETERS. | |
| 9.5. | | |
| 9.6. | | |
| 9.7. | | |
| 9.8. | PHARMACODYNAMIC STATISTICAL ANALYSIS | |
| 10. | INTERIM ANALYSIS | 23 |
| 11. | CHANGES IN THE PLANNED ANALYSIS | 23 |
| 12. | REFERENCES. | 23 |

# **List of Abbreviations**

| List of Abbrevi | <del>-</del> |
|---|---|
| Abbreviation | |
| AE | adverse event |
| ANOVA | analysis of variance |
| AUC | area under the plasma concentration versus time curve |
| $AUC_t$ | area under the plasma concentration versus time curve from time 0 to |
| | the last quantifiable concentration |
| $AUC_{\infty}$ | area under the plasma concentration versus time curve from zero to infinity |
| AUEC | area under the effect versus time curve |
| AUEC <sub>t</sub> | area under the effect versus time curve from time 0 to last quantifiable |
| | concentration time |
| BLQ | below the limit of quantification |
| BMI | body mass index |
| CI | confidence interval |
| CL/F | apparent oral clearance |
| $C_{max}$ | maximum observed plasma concentration |
| CRF | case report form |
| CRU | clinical research unit |
| CTCAE | Common Terminology Criteria for Adverse Events |
| Cu | Copper |
| CV | coefficient of variation |
| EC | enteric-coated |
| ECG | electrocardiogram |
| eDISH | evaluation of drug-induced serious hepatotoxicity |
| E <sub>max</sub> | maximum observed PD concentration in plasma |
| EOS | End of Study |
| ET | early termination |
| FSH | Follicle stimulating hormone |
| GMR | geometric mean ratio |
| ICF | informed consent form |
| MedDRA | Medical Dictionary for Drug Regulatory Activities |
| MSE | mean-square error |
| Mo | molybdenum |
| PBC | primary biliary cholangitis |
| PD | pharmacodynamic |
| PE | physical examination |
| PK | pharmacokinetic(s) |
| PT | preferred term |
| QTcF | QT interval corrected for heart rate using Fridericia's formula |
| RBC | red blood cell |
| SAE | serious adverse event |
| | <u> </u> |

Alexion 

| Abbreviation | Term |
|---|---|
| SAP | statistical analysis plan |
| SD | standard deviation |
| SOC | system organ class |
| TEAE | treatment-emergent adverse event |
| TESAE | treatment-emergent serious adverse event |
| $TE_{max}$ | time to reach maximum observed pharmacodynamic concentration in |
| 1 L <sub>max</sub> | plasma |
| Tlag | time delay between the time of dosing and time of appearance of drug |
| Tag | concentration in plasma |
| $T_{max}$ | time to reach maximum observed concentration in plasma |
| $t_{1/2}$ | terminal elimination half-life |
| V <sub>d</sub> /F | apparent volume of distribution |
| WD | Wilson disease |
| % AUC <sub>extrap</sub> | AUC extrapolated from time t to infinity as a percentage of total AUC |
| $\lambda_{\mathrm{z}}$ | apparent terminal-phase elimination rate constant |

Alexion 

### 1. Introduction

This document outlines the statistical methods to be implemented during the analysis of data collected within the scope of Alexion Pharmaceuticals, Inc., protocol ALXN1840-HV-105 (A Phase 1, Randomized, 2-Period, 2-Sequence, Cross-over Study to Determine the Effect of ALXN1840 on the Metabolism of a CYP2C9 Substrate in Healthy Participants), original version, dated 28 Apr 2020. The purpose of this statistical analysis plan is to define the planned statistical analysis of the study data consistent with the study objectives.

ALXN1840 (bis-choline tetrathiomolybdate; formerly known as WTX101) is a novel, first-in-class, copper (Cu)-protein binding agent in development for the treatment of Wilson disease (WD).

# 2. Objectives

# 2.1. Primary Objective

The primary objective of this study is to determine the effect of ALXN1840 on the pharmacokinetics (PK) of celecoxib, a sensitive CYP2C9 substrate.

# 2.2. Secondary Objective

The secondary objectives of this study are to determine the effect of ALXN1840 on the PK of plasma molybdenum (Mo) with the coadministration of celecoxib and to determine the safety and tolerability of ALXN1840, with the coadministration of celecoxib.

### 3. Investigational Plan

### 3.1. Overall Study Design and Plan

The study is being conducted as a randomized, 2-period, 2-sequence, cross-over study to determine the effect of a single dose of ALXN1840 (perpetrator) on the single dose celecoxib (victim) kinetics in healthy male and female participants.

The study has a Screening period (Day -28 to Day -2), two 11-day study periods (Day 1 to Day 11) with a minimum of 14 days between doses of celecoxib, and an End of Study (EOS) Visit (Day  $15 \pm 2$  days) after Period 2 dosing. Participants will report to the clinical research unit (CRU) on the day prior (Day -1) to both dosing periods.

All participants will receive 1 treatment in each study period; treatment order will be defined based on randomization:

- Treatment A: One 200 mg celecoxib capsule with 240 mL water (fasting).
- Treatment B: One 200 mg celecoxib capsule + 4 × 15 mg ALXN1840 enteric-coated (EC) tablets with 240 mL water (fasting).

Alexion 

Based on randomization, participants will be administered either Treatment A or Treatment B in each period. A wash-out period of at least 14 days must separate dose administration in Period 1 and Period 2. Participants will remain institutionalized from the day prior to dosing until Day 11 following dose administration for each period.

The PK profile of ALXN1840 and celecoxib will be determined by blood sampling following single dose administration over approximately 5 half-lives or more for both study interventions. Blood sampling for PK assessments will occur at pre-dose, 1, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192, 216, 240, and 336 hours post-dose to ensure full assessment of exposure over time. The nominal 336-hour sample for Period 1 is pre-dose sample for Period 2. In addition to PK sampling, safety and tolerability will be assessed by monitoring adverse events (AEs), vital signs, 12-lead electrocardiograms (ECGs), and laboratory parameters.

Following scheduled procedures on Day 11, participants will be discharged from the unit. If there are any participants with clinically significant abnormalities at the time of discharge, the Investigator should notify the Medical Monitor prior to discharge, and participants may be asked to remain institutionalized for further clinical monitoring.

Participants may be asked or required to stay in the CRU between Periods 1 and 2, and/or before the EOS visit, for their own safety, and also to maintain the integrity of the conduct of the study.

The EOS Visit will occur approximately 4 days after discharge from Period 2, after collection of the nominal 336-hour PK sample.

This study will include approximately 38 participants; the overall study population will include a minimum of 40% of each sex.

Participants will be randomized to one of two sequences as described in Table 1.

Table 1: Study design

| Sequence | Treatment Seq | uence | Malea | Female <sup>a</sup> | Total |
|---|---|---|---|---|---|
| Number | Study Period | Study Period | | | |
| | 1 | 2 | | | |
| 1 | A | В | 8 to 11 | 8 to 11 | 19 |
| 2 | В | A | 8 to 11 | 8 to 11 | 19 |
| Total | | | 16 to 22 | 16 to 22 | 38 |

<sup>a</sup>In an effort to achieve balance between males and females in each sequence, there will be no less than 16 and no more than 22 of either sex (ie, a maximum split in either direction of approximately 60%:40%). Randomization will be stratified by sex.

Treatment A -One 200 mg celecoxib capsule with 240 mL water (fasting)

Treatment B – One 200 mg celecoxib capsule  $+4 \times 15$  mg ALXN1840 EC tablets with 240 mL water (fasting)

At the Investigator's discretion, additional participants may be screened to allow for a full enrollment of the study, with a minimum of 40% for each sex. Therefore, it is possible that all eligible participants may not be included. Participants not included in the study will be discharged without dosing on Day 1.

Alexion 

### 3.2. Schema

Figure 1: Study ALXN1840-HV-105 Schematic



Participants will be admitted on Day-1 of each period for Check in procedures. Eligible participants will be randomized on Day 1 immediately prior to dosing in Period 1.

Participants will receive treatment (A or B) based on randomization on Day 1 of each period.

Blood samples for PK analysis of total Mo (as a measure of ALXN1840) and celecox ib will be collected in each period on Day 1 at pre-dose, 1, 2, 3, 4, 5, 6, 8, 12 and 24 hours (Day 2) and then at 24 hour intervals on Days 3, 4, 5, 6, 7, 8, 9, 10, and Day 11. The nominal 336-hour sample for Period 1 will be collected pre-dose in Period 2. Participants will be discharged on Day 11 of each period after completion of all procedures and review of all safety data. The end of study visit (EOS) will occur on Day  $15\pm2$  of Period 2, with the collection of 336-hour PK sample for Period 2.

Participants may be asked or required to stay in the CRU between Periods 1 and 2, and/or before the EOS visit, for their own safety, and also to maintain the integrity of the conduct of the study.

# 3.3. Study Endpoints

### 3.3.1. Primary Endpoints

The primary endpoints include following PK parameters of celecoxib with and without the coadministration of ALXN1840

- C<sub>max</sub>: maximum observed plasma concentration
- AUC<sub>t</sub>: area under the plasma concentration (AUC) versus time curve from time 0 to the last quantifiable concentration
- AUC<sub>∞</sub>: AUC versus time curve from time 0 to infinity

### 3.3.2. Secondary Endpoints

The secondary endpoints include following PK parameters for plasma total Mo with the coadministration of celecoxib and safety assessed parameters

- The PK parameters
  - C<sub>max</sub>
  - AUC<sub>t</sub>
  - AUC<sub>m</sub>

Alexion 

- The safety parameters
  - Incidence of treatment-emergent adverse events (TEAEs) and treatmentemergent serious adverse events (TESAEs)
  - Physical examination (PE)
  - Vital signs measurements
  - Clinical laboratory results
  - 12-lead ECG results

### 4. General Statistical Considerations

All data captured on the case report form (CRF), laboratory safety variables, and PK assessments will be listed on an individual basis by treatment sequence and participant. Summary tables will be presented by treatment and overall, unless otherwise specified.

All pre- and post- dose assessments including repeated and/or unscheduled assessments will be included in the data listing.

Continuous variables will be described using the following descriptive statistics: number of non-missing values (n), arithmetic mean, standard deviation (SD), median, Q1, Q3, IQR, minimum, and maximum, unless otherwise specified. Categorical variables will be summarized using percentages and frequency count.

For the summary statistics of all continuous variables unless otherwise specified, minimum and maximum will be presented to the same number of decimal places as the raw data, mean, median, Q1, Q3, and IQR will be presented to one more decimal places than the raw data, and SD will be presented to two more decimal places than the raw data.

Percentages will be suppressed when the count is zero and will be presented to one decimal place. The denominator for all percentages will be the number of participants in the treatment sequence for the population of interest, unless otherwise specified.

Baseline is defined as the last non-missing assessment (including repeated and unscheduled assessments) prior to treatment on Day 1 (dose day for each period), unless otherwise specified. If there are repeated assessments at a time point, the first non-missing assessment will be included in the summary tables. If the original scheduled measurement at that time point is missing, the next available repeated measurement will be used in the summary tables.

For safety laboratory evaluations, for the purpose of summarization, any numeric values recorded below the lower limit or above the upper limit of quantification will be set to the respective limit for all related summaries. In listings, original results containing inequality sign will be displayed, unless otherwise specified.

Study day will be calculated as follows:

• If assessment date is on or after the dose of treatment, then

Alexion 

Study Day = Assessment Date -Day 1 Date + 1

• Otherwise,

Study Day = Assessment Date – Day 1 Date

All statistical analyses detailed in this statistical analysis plan (SAP) will be conducted using SAS® Version 9.4 or higher (SAS Institute, Inc., Cary, North Carolina) and Phoenix® WinNonlin® Version 8.0 or higher (Certara USA, Inc., Princeton, New Jersey).

# 4.1. Statistical Hypotheses

The primary objective is to determine the effect of ALXN1840 on the PK of celecoxib. There is no formal null hypothesis to be statistically tested and used to drive declaration of study success or failure.

To assure the study has enough participants, to estimate the inhibitory effect of ALXN1840 on the metabolism of celecoxib, the sample size was determined using the conservative 90% confidence interval (CI) and 80% to 125% no-effect boundary approach described in the FDA Guidance "Clinical Drug Interaction Studies —Cytochrome P450 Enzyme- and Transporter-Mediated Drug Interactions" (2020). This guidance notes the 80 to 125% boundaries represent a very conservative standard for drugs that have wide safety "margins" and "the totality of evidence should be taken into consideration when determining the clinical impact of the DDI on the substrate drug". Therefore, if the estimated inhibition effect of ALXN1840 on celecoxib PK lies outside this no-effect boundary, this should not be interpreted as a failed study.

# 4.2. Sample Size

A default of no-effect boundary (80% to 125%) approach will be employed to assess whether there is an inhibition effect on the metabolism of celecoxib in the presence of ALXN1840. For a 2-period crossover study design, assuming the true ratio of the means (celecoxib + ALXN1840 vs celecoxib alone) on the PK parameters is 1 ( $C_{max}$ ; AUC $_{\infty}$ ) and the intra-participant coefficient of variation (CV) is 0.30 (<u>Dennison, 2018</u>), a total sample size of 32 participants can achieve 90% power with two 1-sided tests, each with a type I error rate of 5% (two-sided type I error rate of 10%). The intra-participant CV is estimated using residual mean-square error (MSE) term in the analysis of variance (ANOVA) model. The CV is estimated as  $100\% \times \sqrt{(exp \text{ (MSE)} - 1)}$  for the log-transformed PK parameters. Assuming a 15% dropout rate, approximately 38 participants will be enrolled.

### 4.3. Randomization, Stratification, and Blinding

This is a randomized, open-label, 2-period, 2-sequence, cross-over study. The randomization will be stratified by sex. In an effort to achieve balance between males and females in each sequence, there will be no less than 16 and no more than 22 of either sex (ie, a maximum split in either direction of approximately 60%:40%).

Alexion 

### 4.4. Analysis Set

### 4.4.1. Enrolled Set

The enrolled set will include all participants who sign the informed consent form (ICF).

# 4.4.2. Pharmacokinetic/Pharmacodynamic Analysis Set

The PK analysis set will include all participants who have sufficient plasma samples to have evaluable PK data for celecoxib and/or total Mo (as a measure of ALXN1840) in plasma.

The Pharmacodynamic (PD) analysis set will include all participants who have sufficient plasma samples to have evaluable PD data for total Cu or PUF Cu.

# 4.4.3. Safety Set

The safety set will include all participants who receive at least 1 dose of study intervention.

### 5. Participant Disposition

### 5.1. Disposition

Using the enrolled set, the screen failure of participants will be summarized with counts and percentages by overall. Summary table will include the following:

- Number of participants in the enrolled set (ie, all participants who signed the ICF)
- Number of participants who were screen failures
- Number of participants who were randomized
- Number of participants who failed screen due to COVID-19 related reasons
- Reason for screen failure that was not due to eligibility

Based on the randomized participants, the analysis sets will be summarized with counts and percentages by treatment and overall. Summary table will include the following:

- Number of participants included in PK/PD analysis set
- Reason for exclusion from the PK/PD analysis set
- Number of participants included in safety set
- Reason for exclusion from the safety set

Using the randomized participants, PK analysis set, and safety set respectively, the disposition of participants will be summarized with counts and percentages by treatment and overall. Summary table will include the following:

• Number of participants who completed the study

Alexion 

- Number of participants who discontinued the study
- Reasons for discontinuation
- Number of participants who discontinued the treatment
- Reasons for treatment discontinuation
- Number of participants who were discontinued due to COVID-19

Screen failure data, participant disposition data, and analysis set will be presented in separate data listings for the participants who randomized.

### 5.2. Protocol Deviations

The protocol deviations will be summarized by treatment and overall for the safety set.

All protocol deviations will be presented in a data listing based on randomized participants.

# 6. Demographics and Baseline Characteristics

# 6.1. Demographics and Baseline Characteristics

Age, sex, race, ethnicity, height, and body mass index (BMI) will be collected at Screening; weight will be collected at Screening and Check-in for each period.

Demographic characteristics including age, sex, race, ethnicity, weight (kg), height (cm), and BMI (kg/m²) will be summarized by treatment sequence and overall for the safety set.

Weight measurements collected at Check-in to Dosing Period 1 will be used as baseline for the summary.

Demographic characteristics will be presented in a data listing for the safety set.

# 6.2. Urine Alcohol and Drug screen

Urine alcohol test and urine drug screen will be performed at Screening and Check-in for each period.

Urine alcohol and drug screen results in the safety set will be presented in a data listing for the safety set.

# 6.3. Medical History

Medical history will be collected at Screening.

Medical history results will be presented in a data listing for the safety set with each verbatim term be mapped to a system organ class (SOC) and preferred term (PT) using the Medical Dictionary for Drug Regulatory Activities (MedDRA, Version 23.0 or later).

Alexion 

### 6.4. Inclusion and Exclusion Criteria

Inclusion and exclusion criteria will be confirmed at Screening and Check-in for each period.

Admission criteria deviations are defined as any violation of protocol-defined inclusion/exclusion criteria.

Admission criteria deviations will be presented in a data listing for the participants who randomized.

### 6.5. Genetics

Blood samples for genetic testing of CYP2C9 polymorphism will be collected at clinical Check-in (Day -1) for Period 1.

Genetic testing results will be listed and summarized by treatment sequence and overall for the safety set.

### 7. Treatments and Medications

### 7.1. Prior and Concomitant Medications

Prior medications are defined as medications that were started and ended prior to the first dose of treatment. Concomitant medications are defined as medications that were administered after the first dose of treatment. Medications initiated prior to the first dose of treatment and were continued after the first dose of treatment will be counted as both prior and concomitant medications.

Prior concomitant medications will be summarized by treatment sequence and overall for the safety set. Concomitant medications will be summarized by treatment and overall for the safety set. The anatomical therapeutic chemical code coding scheme of the World Health Organization Drug Dictionary Version March 2019 or later will be used to group medications into relevant categories for the tabulation.

All prior and concomitant medications will be presented in a data listing for the safety set.

### 7.2. Non-Pharmacologic Therapies and Procedures

Non-pharmacologic therapies and procedures will be coded using the MedDRA Version 23.0 or later and will be presented in a data listing for the safety set.

### 7.3. Study Treatments

Study treatments will be administered in each study period at the morning of Day 1 and all participants will receive 1 treatment in each study period. Study treatments are as follow

• Treatment A: One 200 mg celecoxib capsule with 240 mL water (fasting).

Alexion 

• Treatment B: One 200 mg celecoxib capsule  $+4 \times 15$  mg ALXN1840 EC tablets with 240 mL water (fasting).

Any dose of ALXN1840 or celecoxib greater than that specified in the protocol will be considered an overdose.

Study treatment administration data will be presented in a data listing for the safety set.

### 8. Safety Analysis

All safety analyses will be performed on the safety set.

Safety analyses will include an analysis of all AEs, ECGs, clinical laboratory data, physical examinations, and vital sign measurements using descriptive statistics. Summaries will be presented by treatment and overall, unless otherwise stated. Shift tables will be summarized with count and percentages of participants in each category. Percentages will be based on the number of participants with both non-missing baseline and relevant post-baseline results.

No inferential statistical analyses are planned for the safety parameters of this study.

### 8.1. Adverse Events

An AE is any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study intervention.

Adverse events will be analyzed in terms of TEAEs which are defined as any AEs that begin or worsen on or after the first dose of treatment until the EOS or early termination (ET). If the onset date/time of an AE is missing and AE end date is on or after the first dose of treatment, the AE will be defined as treatment-emergent.

All AEs will be listed from the time the participant signs ICF until the EOS or ET Visit.

A treatment-related TEAE is defined as TEAE which was considered to be related to the treatment.

All AEs will be coded by SOC and PT using the MedDRA Version 23.0 or later.

All summary tables will include number and percentage of participants and number of events, unless otherwise stated. For the number of AEs, each occurrence will be counted once. Percentages will be based upon the number of participants in the safety set.

In the summary tables where both SOC and PT are presented, the default ordering of SOC will be alphabetical and the default ordering for PT will be most prevalent (using percentage) PT within each SOC based on Total column. For PTs with the same number of participants, they should be further sorted by number of events and then alphabetically.

Alexion 

In the by-participant analyses, a participant having the same event more than once within the same level of summarization will be counted only once within the same treatment using the most intense or worst highest event (for by toxicity grade summary) or the most related event (for by relationship summary).

In summaries of AEs by treatment, AEs will be summarized according to the most recent treatment received prior to the AE onset, regardless of when the AE ended. For example, an AE that started on or after administration of the treatment on Day 1 in Dosing Period 1 but before the administration of treatment on Day 1 in Dosing Period 2 will be summarized for the treatment in Period 1; an AE that started on or after administration of treatment on Day 1 in Dosing Period 2 will be summarized for the treatment in Period 2. The AEs that started before administration of treatment on Day 1 in Dosing Period 1 will not be summarized unless if the AE meets the TEAE definition, in that case, the AEs will be summarized for the treatment received prior to the AEs worsened.

### 8.1.1. Incidence of Adverse Events

An overview summary of TEAEs will be provided and will include the following

- Participants with at least 1 TEAE
- Participants with at least 1 TEAE related to study drug
- Participants with at least 1 TESAE
- Participants with at least 1 TESAE related to study drug
- Participants who drug withdrawn due to TEAE
- Participants who drug withdrawn due to TEAE related to study drug

The frequency of TEAEs will be tabulated by SOC and PT.

# 8.1.2. Relationship of Adverse Events to Study Drug

The relationship between the study intervention and each occurrence of each AE or SAE is assessed by the Investigator. The relationship will be classified as Related or Not Related.

The frequency of TEAEs will be tabulated by SOC, PT and by relationship.

# 8.1.3. Intensity of Adverse Event

The Investigator will make an assessment of intensity for each AE and SAE reported during the study and assign it to one of the following categories from National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) v5.0, published 27 Nov 2017:

- Grade 1: Mild (awareness of sign or symptom, but easily tolerated)
- Grade 2: Moderate (discomfort sufficient to cause interference with normal activities)

Alexion 

- Grade 3: Severe (incapacitating, with inability to perform normal activities)
- Grade 4: Life-threatening
- Grade 5: Fatal

The frequency of TEAEs will be tabulated by SOC and PT and by intensity.

### 8.1.4. Serious Adverse Events

Serious adverse events (SAEs) will be analyzed in terms of TESAEs which are defined as any SAEs that begin or worsen on or after the first dose of treatment until the EOS or ET.

An SAE is defined as any untoward medical occurrence that at any dose:

- Results in death
- Is life-threatening
- Requires participant hospitalization or prolongation of existing hospitalization
- Results in persistent disability/incapacity
- Is a congenital anomaly or birth defect
- Other situations

The frequency of TESAEs will be tabulated by SOC and PT, and by SOC and PT and by relationship.

Treatment-emergent SAEs will be listed separately.

### 8.1.5. Adverse Events Leading to drug withdrawal

Treatment-emergent AEs leading to drug withdrawal will be listed separately.

# 8.2. Clinical Laboratory Evaluations

Laboratory assessments (including chemistry, hematology, and coagulation) will be performed at Screening, Check-in for each period, Day 2 for each period, Day 5 for each period, Day 10 for each period, and EOS or ET.

Urinalysis will be performed at Screening and Check-in for each period.

Summary statistics and change from baseline for chemistry, hematology, and coagulation will be presented by treatment and by visit. Laboratory parameter values will be graded according to the National Cancer Institute CTCAE. Shift tables will be produced for chemistry, hematology, and coagulation. Shift from baseline grade relative to the reference ranges tables will be presented by treatment and by visit. Shift from changes to the worst highest grade assessed post-dose during the study tables will be presented by treatment. Last recheck values collected prior the dose of treatment will be used as baseline and all rechecks will be deleted from post-dose observations in calculating summary statistics.

Alexion 

All clinical laboratory tests (including chemistry, hematology, coagulation, and urinalysis) will be presented in data listings.

### 8.2.1. Chemistry

Serum chemistry evaluation will include blood urea nitrogen, potassium, bicarbonate, sodium, glucose, aspartate aminotransferase, alanine aminotransferase, chloride, alkaline phosphatase, direct bilirubin, total bilirubin, albumin, creatinine, and creatine phosphokinase.

# 8.2.2. Hematology

Blood hematology evaluation will include platelet count, red blood cell (RBC) count, hemoglobin, hematocrit, RBC indices (including mean corpuscular volume, mean corpuscular hemoglobin, and % reticulocytes), and white blood cell count with differential (including neutrophils, lymphocytes, monocytes, eosinophils, and basophils).

# 8.2.3. Coagulation

Blood coagulation evaluation will include international normalized ratio, partial thromboplastin time, and prothrombin time.

# 8.2.4. Urinalysis

Urinalysis evaluation will include specific gravity, pH, glucose, protein, blood, bilirubin, urobilinogen, nitrite, leukocyte esterase by dipstick, and microscopic examination.

### 8.3. Vital Sign Measurements

Oral temperature, pulse rate, respiratory rate, and systolic and diastolic blood pressure (mm Hg) will be performed at Screening, Day 1 (Pre-dose, 1 Hour, 4 Hour, 8 Hour, and 12 Hour) for each period, Day 2 (24 Hour) for each period, and EOS or ET.

Weight will be collected at Screening and Check-in for each period. BMI will be collected at Screening only.

Blood pressure and pulse measurements should be preceded by at least 5 minutes of rest for the participant in a quiet setting without distractions (eg, television, cell phones).

Summary statistics and change from baseline for vital signs (temperature, pulse rate, respiratory rate, and systolic and diastolic blood pressure) will be presented by treatment and overall and by visit and time point. Last recheck values collected prior to the dose of treatment will be as baseline and all rechecks will be deleted from post-dose observations in calculating summary statistics.

Vital sign measurement results, including height, weight, and BMI, will be presented in a data listing.

Alexion 

### 8.4. Physical Examination

A full PE, at a minimum, assessments of the cardiovascular, respiratory, gastrointestinal, and neurological systems will be performed at Screening, Check-in for each period, and EOS or ET. A symptom-driven physical examination may be performed at other times, at the principal investigator's discretion.

General appearance, skin, head/ear/eye/nose/throat, neck, lymph node, chest, heart, abdominal cavity, limb, central nervous system, and musculoskeletal will be captured on the CRF.

Physical examination results will be presented in a data listing.

### 8.5. Electrocardiogram

Triplicate 12-lead ECG will be performed at Screening and Day 1 (Pre-dose and 4 Hour [before lunch]) for each period.

Participants will be resting in the supine position for at least 15 minutes prior to and 5 minutes after each nominal time point for ECG extraction.

Heart rate, PR interval, QRS interval, RR interval, QT interval, QT interval corrected for heart rate using Fridericia's formula (QTcF), and interpretation of ECG will be captured on the CRF.

The average of the triplicate ECG readings at the time points collected will be calculated. Summary statistics and change from baseline of calculated average for heart rate, PR interval, QRS interval, RR interval, QT interval, and QTcF interval will be presented by time point. Last recheck values collected prior to the dose of treatment will be as baseline and all rechecks will be deleted from post-dose observations in calculating summary statistics.

Triplicate 12-lead ECG findings will be presented in a data listing.

# 8.6. Other Safety Data

### 8.6.1. Liver Function Results

All events of ALT  $\geq$  3 × upper limit of normal (ULN) and bilirubin  $\geq$  2 × ULN ( $\geq$  35% direct bilirubin) or ALT  $\geq$  3 × ULN and international normalized ratio (INR)  $\geq$  1.5, if INR measured which may indicate severe liver injury (possible Hy's Law), must be reported as an SAE (excluding studies of hepatic impairment or cirrhosis).

Liver function results will be presented in a summary table and eDISH (evaluation of drug-induced serious hepatotoxicity) plots.

# 8.6.2. Serology

Serology including HIV, hepatitis B, and hepatitis C screen will be performed at Screening.

Alexion 

Serology results will be presented in a data listing.

### 8.6.3. Pregnancy Test

Serum or urine pregnancy test for female participants and female spouses/partners of male participant will be performed at Screening, Check-in for each period, and EOS or ET.

Pregnancy test results will be presented in a data listing.

# 8.6.4. Follicle Stimulating Hormone

Follicle stimulating hormone (FSH) will be performed at Screening and only needed if claiming exemption from contraception requirement due to menopause.

FSH results will be presented in a data listing.

### 8.6.5. Discussion/documentation of contraception method

Discussion/documentation of contraception method will be performed at Screening and Check-in for each period. The discussion/documentation of contraception method results will be kept in the source documents and will not be recorded on the CRF; therefore, the discussion/documentation of contraception method results will not be presented in any of the tables, listings, or figures.

# 8.6.6. Retained Sample

A single 12 mL sample will be retained for evaluation in the event of an unexpected safety finding; retained samples may be destroyed after completion of the clinical study report. The retained serum sample will only be collected pre-dose on Day 1 of Period 1.

Retained sampling results will be presented in a data listing.

### 9. Pharmacokinetics and Pharmacodynamic Analysis

### 9.1. Pharmacokinetic Sampling

Whole blood samples will be collected for the measurement of plasma concentrations of total Mo, PUF Mo, and celecoxib at the following time points: pre-dose and post-dose at 1, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192, 216, 240, and 336 hours in each period. Additional samples may be collected at additional time points during the study if warranted and agreed upon between the Investigator and Alexion. Collection of samples for PK evaluation should occur as close as possible to the scheduled time and actual time of collection should be documented on the eCRF. Samples collected within  $\pm$  10% of the scheduled time, or 30 minutes, whichever is less, will not be considered a protocol deviation. In the event of a safety occurrence and after agreement between the Investigator and Medical Monitor, up to 3 additional PK sampling timepoints may be added.

PK samples will also be used for the PD analysis of total Cu and PUF Cu.

Alexion 

# 9.2. BLQ Values / Missing Values

For PK and the PD measure Total Cu parameter calculations, concentrations below the limit of quantification (BLQ) prior to the first measurable concentration will be set to zero; all other BLQ values will be treated as missing. For PUF Cu parameter calculations, all BLQ values will be set to zero.

For PK and PD concentration summaries, BLQ values will be set to zero.

# 9.3. Pharmacokinetic/Pharmacodynamic Data Presentation Conventions

PK and PD concentration data will be summarized using descriptive statistics (number of participants (N), number of participants with available data (n), arithmetic mean, SD, arithmetic CV, geometric mean (GM), geometric CV, median, minimum and maximum).

The predose PD concentration will be used as baseline; absolute change from baseline will be calculated as: a postdose concentration value – baseline concentration value; percent change from baseline will be calculated as: ([a postdose concentration value – baseline concentration value] / baseline) ×100%.

The following conventions will be applied to PK/PD presentations and summaries.

- For continuous variables, all mean and median values are formatted to one more
  decimal place than the measured value. Standard deviation values are formatted to
  two more decimal places than the measured value. Minimum and maximum
  values are presented with the same number of decimal places as the measured
  value.
- Date variables are formatted as DDMMMYYYY for presentation. Time is formatted in military time as HH:MM for presentation.

### 9.4. Pharmacokinetic Parameters

The following plasma PK parameters will be calculated for total Mo, PUF Mo, and celecoxib using noncompartmental methods with Phoenix® WinNonlin® (Certara USA Inc., Princeton, New Jersey) Version 8.0 or higher or SAS Version 9.4 or higher (SAS Institute Inc., Cary, North Carolina), as applicable. Calculations will be based on the actual sampling times relative to the actual reference ALXN1840 dosing times recorded during the study.

- T<sub>lag</sub>: time delay between the time of dosing and time of appearance of drug concentration in plasma (for plasma total Mo and PUF Mo with ALXN1840 administration)
- C<sub>max</sub>: maximum observed concentration in plasma
- T<sub>max</sub>: time to reach maximum observed concentration in plasma
- AUC<sub>t</sub>: AUC from time 0 to the last quantifiable concentration, calculated using the linear trapezoidal rule

Alexion 

- AUC $_{\infty}$ : AUC versus time curve from time 0 to infinity, calculated using the linear trapezoidal rule
- % AUC extrapolated from time t to infinity as a percentage of total AUC  $_{\infty}$
- $t_{1/2}$ : terminal elimination half-life
- $\lambda_z$ : apparent terminal-phase elimination rate constant

For ALXN1840, equivalent Mo dose will be used to calculate total Mo (and PUF Mo if applicable) CL/F and Vd/F values: Mo MW of 95.95 Da/ALXN1840 MW of 432.54 Da x 60 mg ALXN1840 = 13.31 mg Mo dose. For celecoxib, use 200 mg dose for the calculation.

- CL/F: apparent oral clearance
- V<sub>d</sub>/F: apparent volume of distribution

Additional plasma PK parameters may be calculated if deemed appropriate.

### 9.5. Pharmacokinetic Statistical Analysis

Plasma concentration data for total Mo, PUF Mo, and celecoxib will be summarized separately for each scheduled sampling time using descriptive statistics. Plasma concentrations of total Mo, PUF Mo, and celecoxib and time deviation data will be presented in a data listing by participant. Mean plasma concentration versus scheduled time profiles will be presented in figures on both linear and semilogarithmic scales. Individual plasma concentration versus actual time profiles will be presented similarly.

Pharmacokinetic parameters derived from plasma concentrations of total Mo, PUF Mo, and celecoxib will be presented in data listings and summarized separately using the following descriptive statistics: N, n, arithmetic mean, SD, arithmetic CV, median, minimum, maximum, and 95% confidence interval (CI). Geometric mean and geometric CV will be presented for  $C_{max}$  and AUCs only.

The effect of ALXN1840 on celecoxib PK will be assessed using a linear mixed-effect model (SAS PROC MIXED) with treatment condition, sequence, and period as fixed effects and participant nested within sequence as a random effect. The model will be fitted to the natural-log-transformed PK parameters  $C_{max}$ ,  $AUC_{\infty}$  and  $AUC_{t}$  for estimation of effects and construction of CIs for the test treatment (Treatment B: 200 mg celecoxib + 60 mg ALXN1840) compared with the reference treatment (Treatment A: 200 mg celecoxib). The within-participant CV for the corresponding PK parameters will be estimated using the mean squared error from the statistical model. Confidence intervals (90%) will be constructed for the least-squares geometric mean ratio (GMR) estimates between the test and reference treatments for the indicated PK parameters using the natural log-transformed data. The GMR estimates and the associated 90% confidence limits will

Alexion 

be exponentiated back to the original scale. The statistical results will also be graphically presented using a forest plot.

# 9.6. Genetic Variant Analyses for CYP2C9

Participants with variant CYP2C9 alleles will be identified in the PK concentration and parameter listings, where applicable. The characterization of potential impact of ALXN1840 on phenotypic CYP2C9 metabolism of celecoxib and genetic polymorphism on the between-participant variability of celecoxib PK are exploratory assessments. Thus, this study does not specifically select target participants with a certain proportion of CYP2C9 genotypes. Depending on the distribution of CYP2C9 genotypes within treatments, the impact of ALXN1840 coadministration on celecoxib PK may be stratified by CYP2C9 genotypes to assess the impact on the drug-drug interaction.

### 9.7. Pharmacodynamic Parameters

The following plasma PD parameters will be calculated using noncompartmental methods for Total Cu and PUF Cu (measured and absolute change from baseline) concentrations with Phoenix® WinNonlin® (Certara USA Inc., Princeton, New Jersey) Version 8.0 or higher or SAS Version 9.4 or higher (SAS Institute Inc., Cary, North Carolina), as applicable. Calculations will be based on the actual sampling times relative to the actual reference ALXN1840 dosing times recorded during the study.

- E<sub>max</sub>: maximum observed PD concentration in plasma
- TE<sub>max</sub>: time to reach maximum observed PD concentration in plasma
- AUEC<sub>t</sub>: area under the effect versus time curve (AUEC) from time 0 to last quantifiable concentration time, calculated using the linear trapezoidal rule

Additional PD parameters may be calculated as necessary.

### 9.8. Pharmacodynamic Statistical Analysis

Plasma concentration data for total Cu and PUF Cu will be summarized separately for each scheduled sampling time using descriptive statistics. Individual concentration data will be presented in data listings. Individual concentration versus actual time profiles will be provided. Additionally, mean concentration versus nominal time profiles will be provided. Note that the measured, change from baseline, and percent change from baseline concentration data for total Cu and PUF Cu will be listed, summarized, and presented graphically on linear scales.

Parameters for total Cu and PUF Cu in plasma will be summarized separately using descriptive statistics (N, n, mean, SD, median, %CV, minimum, and maximum). Geometric mean and geometric %CV will be calculated for AUECs and  $E_{max}$ .

Alexion 

# 10. Interim Analysis

No interim analyses are planned for this study.

# 11. Changes in the Planned Analysis

For the definition of PK/PD analysis set in the protocol was "All participants who have sufficient plasma samples to have evaluable PK data for celecoxib and total Mo (as a measure of ALXN1840) in plasma", in this SAP is changed to "The PK analysis set will include all participants who have sufficient plasma samples to have evaluable PK data for celecoxib and/or total Mo (as a measure of ALXN1840) in plasma. The Pharmacodynamic (PD) analysis set will include all participants who have sufficient plasma samples to have evaluable PD data for total Cu or PUF Cu."

### 12. References

Dennison J, Puri A, Warrington S, Endo T, Adeloye T, Johnston A. Amenamevir: Studies of Potential CYP2C8- and CYP2B6-Mediated Pharmacokinetic Interactions With Montelukast and Bupropion in Healthy Volunteers. Clin Pharmacol Drug Dev. 2018;7(8):860-870.

Alexion 



# **PPD Biostatistics and Programming**

Statistical Analysis Plan (SAP) Client Approval Form

| Client: | Alexion Pharmaceuticals, Inc. |
|---|---|
| Protocol Number: | ALXN1840-HV-105 |
| Document Description: | Final Statistical Analysis Plan |
| SAP Title: | A Phase 1, Randomized, 2-Period, 2-Sequence,<br>Cross-over Study to Determine the Effect of ALXN1840<br>on the Metabolism of a CYP2C9 Substrate in Healthy<br>Participants |
| SAP Version Number: | Version 1.0 |
| Effective Date: | 04 Sep 2020 |

# Author(s): For PPD: PPD For PPD: PPD



PPD CONFIDENTIAL AND PROPRIETARY

| mmm° | PPD Biostatis | stics and Programming | |
|---|---|---|---|
| <i>PPU</i> | Statistical Analysis Plan (S. | AP) Client Approval Form | |
| | PPD | 04-Sep-2020 14:23:05 | EDT |
| PPD PPD | | Date (DD-MMM-YYYY) | |
| Alexion Pharmace | | | |

SOP-BST-05ar06 Effective Date: 19 September 2019 Page 2 of 2



# **Certificate Of Completion**

Envelope Id: PPD

Subject: Please DocuSign: ALXN1840-HV-105 SAP Approval Form.pdf

Source Envelope:

Document Pages: 2 Certificate Pages: 2

AutoNav: Enabled
Envelopeld Stamping: Disabled

Time Zone: (UTC-05:00) Eastern Time (US & Canada)

Status: Completed

Envelope Originator:

PPD

100 College St.

New Haven, CT 06510

PPD

IP Address: PPD

### **Record Tracking**

Status: Original

04-Sep-2020 | 12:47

Holder: PPD

Signatures: 4

Initials: 0

Location: DocuSign

**Timestamp** 

Sent: 04-Sep-2020 | 13:35

Viewed: 04-Sep-2020 | 13:51

Signed: 04-Sep-2020 | 13:51

Sent: 04-Sep-2020 | 13:35

Viewed: 04-Sep-2020 | 13:35 Signed: 04-Sep-2020 | 13:36

### **Signer Events**

PPD

PPD

PPD

Alexion Pharmaceuticals, Inc.

Security Level: Email, Account Authentication

(Required)

Signature

PPD

PPD

Signature Adoption: Pre-selected Style

Signature ID:

PPD

Using IP Address: PPD

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I approve this document

# **Electronic Record and Signature Disclosure:**

Not Offered via DocuSign

PPD PPD

PPD

Alexion Pharmaceuticals Inc.

Security Level: Email, Account Authentication

(Required)

PPD

Signature Adoption: Pre-selected Style

Signature ID:

PPD

Using IP Address: PPD

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I approve this document

**Electronic Record and Signature Disclosure:** 

Not Offered via DocuSign

**Signer Events Signature Timestamp** PPD Sent: 04-Sep-2020 | 13:35 PPD PPD Viewed: 08-Sep-2020 | 07:10 PPD Signed: 08-Sep-2020 | 07:11 Alexion Pharmaceuticals, Inc. Signature Adoption: Pre-selected Style Security Level: Email, Account Authentication Signature ID: (Required) PPD Using IP Address: PPD With Signing Authentication via DocuSign password With Signing Reasons (on each tab): I approve this document **Electronic Record and Signature Disclosure:** Not Offered via DocuSign PPD PPD Sent: 04-Sep-2020 | 13:35 PPD Viewed: 04-Sep-2020 | 14:22 Signed: 04-Sep-2020 | 14:23 Alexion Pharmaceuticals, Inc. (Regulated) Signature Adoption: Pre-selected Style Security Level: Email, Account Authentication Signature ID: (Required) PPD Using IP Address: PPD With Signing Authentication via DocuSign password With Signing Reasons (on each tab): I approve this document **Electronic Record and Signature Disclosure:** Not Offered via DocuSign

| In Person Signer Events | Signature | Timestamp |
|---|---|---|
| Editor Delivery Events | Status | Timestamp |
| Agent Delivery Events | Status | Timestamp |
| Intermediary Delivery Events | Status | Timestamp |
| Certified Delivery Events | Status | Timestamp |
| Carbon Copy Events | Status | Timestamp |
| , , | | |
| Witness Events | Signature | Timestamp |
| | Signature<br>Signature | Timestamp Timestamp |
| Witness Events | _ | · |
| Witness Events Notary Events | Signature | Timestamp |
| Witness Events Notary Events Envelope Summary Events | Signature<br>Status | Timestamps |
| Witness Events Notary Events Envelope Summary Events Envelope Sent | Signature Status Hashed/Encrypted | Timestamps 04-Sep-2020 13:35 |
| Witness Events Notary Events Envelope Summary Events Envelope Sent Certified Delivered | Status Hashed/Encrypted Security Checked | Timestamps 04-Sep-2020 13:35 08-Sep-2020 07:10 |